CLINICAL TRIAL: NCT03951246
Title: The Effect of Cognitive and Motor Training on Executive Functions, Motor Skills, and Saccadic Eye Movements System in Pediatric Posterior Fossa Tumor Survivors
Brief Title: Cognitive and Motor Training in Pediatric Posterior Fossa Tumor Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal Research Institute of Pediatric Hematology, Oncology and Immunology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 8э/15-17
Record Dates: First submitted 2019-02-13; First posted 2019-05-15 (Actual); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Childhood Cancer; Cognitive Impairment; Motor Skills Disorders; Posterior Fossa Tumor
Keywords: executive functions; motor skills; eye tracking; pediatric cancer; posterior fossa tumors
MeSH Terms: conditions — Neoplasms; Cognitive Dysfunction; Motor Skills Disorders; Infratentorial Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training Group (Experimental): Training Group recieved cognitive and Motor training included 6 sessions using the following training devices.
  * Dynavision D2 ® (USA) (https://products.dynavisioninternational.com/products/d2) presents a panel with 64 bulbs which take the form of five circles. The task of a participant is to press the bulb that is glowing as quick as possible. In the trial 8 modes will be used; they have different instructions which are aimed at visual-motor co-ordination, processing speed, inhibition, and shifting.
  * Fitlight Trainer ® (Canada) (https://www.fitlighttraining.com) consists of 7 clickers, and the tasks are similar to Dynavision ones.
  * NeuroTracker ® (Canada) (https://neurotracker.net) includes a task of multiple object training for working memory and attention enhancement.
  Interventions: Other: Cognitive and Motor Training
- Control Group (No Intervention): Control Group didn't recieved any cognitive and motor training. They visited swimming pool and physical therapy.

INTERVENTIONS:
Other: Cognitive and Motor Training — In the first phase of the trial, all participants (patients and healthy children) will complete cognitive and motor functions assessment.
  Then the sample of patients who have cognitive/motor impairment will be randomized to an either Intervention or Control group.
  In the second phase of the trial, survivors in the Intervention Group will receive 6 sessions of cognitive and motor training during two weeks, and survivors in Control Group will undergo …..
  After this treatment phase, motor and cognitive functions assessment will be conducted in all patients once again.
  In the third phase, the Control Group will be provided the active intervention (i.e. 6 sessions of cognitive and motor training during two weeks), while the Intervention Group engages in passive reading.
  After this, motor and cognitive functions assessment will be carried out in all patients once again.
  Arms: Training Group

SUMMARY:
The purpose of this study is to create a rehabilitation program for children who survived posterior fossa tumors using the latest technology. Supposed that training in Fitlight, Dynavision D2, NeuroTracker will improve executive functions, visual-motor integration, fine and gross motor functions.

DETAILED DESCRIPTION:
The death rates from posterior fossa tumors (PFT) have declined significantly over the past decades. Children and adolescents who survived this kind of tumor without metastases demonstrate 5-year survival rates of 90%. Standard treatment for posterior fossa tumors includes surgical rejection, which can be combined with radiotherapy and chemotherapy. However, treatment factors can cause the impairment of motor and cognitive functions, which influence negatively speech, academic achievements, and quality of life. Such an outcome can be induced by tumor growth process as well. One of the most essential consequences of the disease is cognitive deficiency in the areas of attention, working memory, and executive functions.

The cerebellum pathology often causes deficits of motor skills. Considering that motor system has a hierarchal organization, PFT can cause the impairment of all the system, starting with gross motor skills and ending in the finest eye movements. The cerebellum has been shown to control voluntary eye movements, particularly such parameters as accuracy and velocity of saccades, fixation duration, etc.

Given the effect of probable deficits on a child's daily life, the issue of cognitive and motor remediation programs is in the spotlight today. There is some evidence that interventions targeting cognitive functions (e.g. working memory, short-term memory, attention, planning) and motor skills (gross and fine motor skills, muscle strength, agility) can be effective in these patients.

However, only few of remediation programs focus on visual-motor co-ordination and saccadic eye movements system, despite the fact that they provide the basis for higher-level functions, such as sustained attention, working memory, and planning.

The research conducted in Clinical Rehabilitation Research Center "Russkoe Pole" has revealed that treatment gains in the areas of motor skills, and specifically saccadic eye movements, are positively associated with the enhancement of attention and working memory. Given this, the investigators can suggest that this improvement is connected with the reduction of extra saccadic movements and consequently the decrease of irrelevant information to be processed. This mechanism can be generalized to the other executive functions, such as shifting, inhibition, and planning.

This trial will allow the investigators to determine potential feasibility of rehabilitation program targeting motor and cognitive functions, as well as the saccadic system, in pediatric posterior fossa tumor survivors.

ELIGIBILITY:
Inclusion Criteria:

* Survivor of posterior fossa tumor/healthy control
* Currently aged 6-17
* Staying in Clinical Rehabilitation Research Center for 32 days
* Research participant or legal guardian/representative to give written informed consent

Exclusion Criteria:

* Currently on stimulants or other medications intended to treat motor or cognitive impairment
* History of seizures
* Severe deficits in vision, motor skills, or cognitive functions
* Inability or unwillingness of research participant or legal guardian/representative to give written informed consent

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-05-21 (Actual); Study Completion 2018-05-21 (Actual)

PRIMARY OUTCOMES:
Eye tracking | Change from Baseline Eye tracking mesuares up to 2 weeks and follow-up after 4 weeks from Baseline
  Following outcomes are mesuared: Execution time, Number of Fixations, Scan Path, Mean Duration of Fixations, Mean Saccades Amplitude, Ellipse Square
VMI | Change from Baseline VMI mesuares up to 2 weeks and follow-up after 4 weeks from Baseline
  Following outcomes are mesuared: Visual-motor integration, Visual perception, Motor coordination.
Dynavision | Change from Baseline Dynavision mesuare up to 2 weeks and follow-up after 4 weeks from Baseline
  Following outcome are mesuared: Reaction Time
Fitlight | Change from Baseline Fitlight mesuare up to 2 weeks and follow-up after 4 weeks from Baseline
  Following outcome are mesuared: Reaction Time
Neurotracker | Change from Baseline Neurotracker mesuare up to 2 weeks and follow-up after 4 weeks from Baseline
  Following outcome are mesuared: Score
CANTAB | Change from Baseline CANTAB mesuare up to 2 weeks and follow-up after 4 weeks from Baseline
  Following outcomes are mesuared: Pattern Recognition Memory Immediate, Pattern Recognition Memory Delayed, Spatial Recognition Memory, Spatial Working Memory (Mistakes), Spatial Working Memory (Strategy), Spatial Span, Rapid Visual Processing (Mistakes), Rapid Visual Processing (Median Latency)
BOT-2 | Change from Baseline BOT-2 mesuare up to 2 weeks and follow-up after 4 weeks from Baseline
  Following outcomes are mesuared: Fine Motor Skills, Gross Motor Skills, Coordination, Strength and Agility, General Score

CONTACTS AND LOCATIONS:
Locations (1):
- Dmitry Rogachev Federal Research and Clinical Centre of Paediatric Haematology, Oncology and Immunology, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No
The software product, within which the interaction between patients and specialists will be realized, is supposed to be created in the Splunk system. The system allows to search both the real-time data and the archived data, based on the results of the search Splunk gives you the opportunity to: analyze the results with the visualization tools, generate reports and warnings, create a monitoring and notification systems in real time. These can be expanded - you can create new applications using the specialized development platform that comes with Splunk. The study will be attended by at least 1000 patients and their families who have concluded an agreement with the Medical-Rehabilitation Scientific Center "Russe pole", and come to the examination at least 2 times a year.